CLINICAL TRIAL: NCT05832463
Title: Effects of a Novel Carbohydrate Blocking Supplement on Glycemic Variability as Measured by Continuous Glucose Monitoring
Brief Title: Effects of a Novel Supplement on Glycemic Variability Measured by Continuous Glucose Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dōTERRA International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: DO-120043-CBS
Record Dates: First submitted 2023-03-10; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Carbohydrate blocking supplement; Continuous Glucose Monitoring; Interstitial glucose levels

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 1 is single-blind. Participants will not know their treatment allocation in either arm of the study. Furthermore, in cohort 1, the participants may receive a 250 mg or 500 mg CBS dose, but will not be informed which they receive. In order to preserve blinding to dosage allocation, participants will be instructed to consume two capsules prior to each meal.
  * Participants receiving the 500 mg CBS dose will take 2 CBS capsules
  * Participants receiving the 250 mg CBS dose will take 1 CBS capsule and 1 placebo capsule
  * Participants in the placebo arm will take 2 placebo capsules
  Cohort 2 is double blind - participants will know that they will receive either the treatment or placebo first, but will be blinded to which they receive. All members of research staff will be blinded with the exception of a designated member
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): In cohort 1, participants will receive either a 250 mg mulberry leaf extract CBS dose (1 supplement capsule t.i.d. + 1 placebo capsule to preserve blinding) or a 500 mg mulberry leaf extract CBS dose (2 supplements t.i.d.) in the experimental arm and will cross over to or from the placebo arm.
  In cohort 2, participants will receive a 500 mg mulberry leaf extract CBS dose (2 supplement capsules t.i.d.) in the experimental arm and will cross over to or from the placebo arm.
  Interventions: Dietary Supplement: Carbohydrate blocking supplement (CBS)
- Placebo arm (Placebo Comparator): In Cohorts 1 and 2, participants will receive 2 placebo capsules in the placebo arm and will cross over to or from the experimental arm.
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Carbohydrate blocking supplement (CBS) — The CBS is composed of a Hypromellose outer shell, and filled with mulberry leaf extract, berberine HCl, cinnamon bark powder, and cinnamon bark essential oil.
  Mulberry leaf extract (Reducose) - 250 mg Berberine HCl (97%)(Berberis aristata root extract)- 25 mg Organic cinnamon powder (Cinnamon (Cinnamomum loureirii) bark powder) - 20 mg Essential oil blend (Grapefruit (Citrus paradisii) peel oil, Lemon (Citrus limon) peel oil Peppermint (Mentha piperita) aerial (leaf/stem) oil), Ginger (Zingiber officinale) root oil, Cinnamon (Cinnamomum zeylanicum) bark oil) - 5 mg
  Arms: Experimental arm
Dietary Supplement: Placebo capsule — The placebo is composed of a Hypromellose outer shell filled with extra virgin olive oil.
  Arms: Placebo arm

SUMMARY:
This is a two-cohort, crossover pilot study to determine interstitial glucose levels coincident with the consumption of a novel carbohydrate blocking supplement.

DETAILED DESCRIPTION:
This two-cohort study will evaluate a novel supplement developed for metabolic support using measures of glycemic variability, fasting glucose, and fasting insulin. In the first cohort, over the course of two weeks, these endpoints will be determined by continuous glucose monitoring (CGM) and blood/urine analyses in healthy adults using a carbohydrate blocking supplement (CBS). Following an interim analysis, the CBS will be evaluated for an additional two months in healthy volunteers using the same measures outlined above.

ELIGIBILITY:
Inclusion Criteria:

If female, negative pregnancy test

* Body mass index (BMI) ≤ 32
* HbA1C ≤ 6.4% at screening
* Fasting blood glucose level ≤ 125 mg/dL at screening
* [COHORT 1 ONLY] Willing and able (in the opinion of the investigator) to comply with all study requirements, including swallowing size 00 capsules (approximately 23 mm long and 8.5 mm diameter), food journaling, consumption of a standardized, high carbohydrate meal daily, CGM device application, and phlebotomy
* [COHORT 2 ONLY] Willing and able (in the opinion of the investigator) to comply with all study requirements, including swallowing size 00 capsules (approximately 23 mm long and 8.5 mm diameter), CGM device application, and phlebotomy
* Signed informed consent, HIPAA Authorization, and Confidentiality Agreement

Exclusion Criteria:

* Pregnancy within the last 60 days or currently breastfeeding
* Existence of any medical condition, significant disease or disorder, or surgery within the past 12 months that may, in the judgment of the medical provider, put the participant at risk, or affect study results, procedures or outcomes
* Existence of any medical concerns, or any finding that may, in the judgment of the staff medical provider, put the participant at risk, or affect study results, procedures or outcome
* [COHORT 1 ONLY] Sensitivity or allergy to gluten, sugar, peanuts, apples, strawberries, dairy, or orange juice
* Known or suspected allergy or sensitivity to essential oil, fatty oils, cellulose, or botanical products
* Currently following a ketogenic or medically prescribed diet, or have followed a ketogenic or medically prescribed diet within the last 3 months
* Arterial hypertension ≥140/90 mmHg.
* HbA1c ≥ 6.5% at screening
* Fasting blood glucose > 125 mg/dL at screening
* Current or previous participation in any other clinical trial within the last month
* History of smoking or vaping within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability (cohort 1) | 2 weeks
  This study will monitor the occurrence and frequency of adverse events and safety, both through participant report and blood chemistry/hematology analyses. Dosage for cohort 2 will be determined
Dose determination for Cohort 2 | 2 weeks
  Dosage for cohort 2 will be determined
Glucose levels monitoring (Cohort 2) | 2 months
  Use of continuous glucose monitoring (CGM) to monitor interstitial glucose levels
Glycemic variability (Cohort 2) | 2 months
  Glycemic variability will be determined in healthy individuals.

SECONDARY OUTCOMES:
Glucose levels monitoring (Cohort 1) | 2 weeks
  Use of continuous glucose monitoring (CGM) to monitor interstitial glucose levels
Glycemic variability (Cohort 1) | 2 weeks
  Use of continuous glucose monitoring (CGM) to monitor interstitial glucose levels and Glycemic variability will be determined in healthy individuals.
Albumin (g/dL) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
BUN (mg/dL) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Creatinine (mg/dL) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Alkaline phosphatase (U/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
ALT (U/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
AST (U/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Calcium (mg/dL) | 2 weeks, 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Carbon Dioxide (mmol/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Chloride (mmol/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Potassium (mmol/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Sodium (mmol/L) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Total bilirubin (mg/dL) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Total protein (g/dL) | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Item in comprehensive metabolic panel for safety assessment
Fasting insulin | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Fasting insulin to determine changes, if any, to metabolism.
Fasting glucose | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Fasting glucose to determine changes, if any, to metabolism.
Body weight | 2 weeks (Cohort 1), 2 months (Cohort 2)
  Determine whether body weight is affected by the consumption of the study product.
Safety/tolerability (cohort 2) | 2 months
  This study will monitor the occurrence and frequency of adverse events and safety, both through participant report and blood chemistry/hematology analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Osguthorpe, MD, Principal Investigator — doTERRA International
Locations (1):
- doTERRA International, Pleasant Grove, Utah, United States